CLINICAL TRIAL: NCT03394313
Title: Qatar Cardiometabolic Registry
Status: Recruiting | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-17-003
Record Dates: First submitted 2018-01-01; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
Keywords: Registry
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD) are closely related. T2DM risk equivalent for CVD and it remains the major cause of death in T2DM. Thus, patients with T2DM and CVD disease are at very high-risk of CVD-related mortality. Therefore, more aggressive metabolic and hemodynamic control is required in such patients to improve the prognosis. We recently initiated a cardio-metabolic clinical service at the Heart Hospital, where T2DM patients with existing CVD are simultaneously examined by Cardiologist and Diabetologist for optimal metabolic and hemodynamic control. We would like to start a clinical registry for all patients who attend this clinical service to collect import clinical data about this population. This registry will serve an important source for future clinical research in the field.

DETAILED DESCRIPTION:
Various investigators have shown that type 2 diabetes is associated with out-of-hospital cardiac arrest and mortality due sudden cardiac arrest [1,2]. In comparison to non-diabetic patients, those with T2DM possess greater risk of cardiovascular morbidity and deaths, and are considerably influenced by cardiovascular disease [3]. To assess the potential benefit of T2DM prevention and treatment, as well as the future burden of T2DM-associated diseases can help in better understanding of the T2DM and the risk of chronic cardiovascular manifestations is warranted [4]. Herein, we would like to start a clinical registry for all patients who attend this clinical service to collect import clinical data about this population. This registry will serve an important source for scientific information that can be used in future to design clinical research studies for better patient care and management.

The cardio-metabolic clinic has been recently established in the Heart Hospital to provide state-of-the-art care for patients with T2DM and established heart disease, e.g. ischemic heart disease, heart failure, etc. the health information of all patients attending the cardio-metabolic Clinic for the care of their disease who provide their consent for the use of their health information in the registry will be added to the registry.

A data base for this registry will be created in Cerner which will be password protected. Clinical information about patients attending the cardiometabolic clinic in the Heart Hospital will be collected. Data will include demographics (age, gender, and nationality), vital signs (Pulse rate, blood pressure), waist circumference , Weight, Canadian Cardiovascular Society (CCS) Class, New York Heart Association ( NYHA) class, history of hospitalization for chest pain, shortness of death, Stent thrombosis, syncope or Dizzy spells, Stroke, Transient Ischemic Attack (TIA), Polyurea, urinary tract infection, Activity Level, Foot exam, Peripheral pulses, Mono-filament exam, Ankle Brachial Index test, Cardiac Rehabilitation, Diabetes monitoring at home, Insulin Pump, Revascularization Needed, angiogram and presentation (Presenting Acute Coronary Syndrome (ACS), ST-Elevation Myocardial Infarction (STEMI), Upstream antiplatelets, Culprit artery, Non-ST-Elevation Myocardial Infarction (NSTEMI), Stent-No1, Unstable angina, Known Diabetes, Stent-No2, Newly diagnosed DM, Stent-No3, Hypertension, Total No of Stent, Tobacco use, Type of Stent, Thrombectomy, Troponin highest level, EUROScore, Reopro, Coronary angiogram, Thrombosis in Myocardial Infarction (TIMI) flow, Dissection, Perforation, Syntax Score Coronary Artery Disease (SYNTAXSCORE), Left Main Coronary Artery (LM), Loss of side branch, Access type, Left Anteriour Descending Artery (LAD), D1, Seal Device, D2, Left Circumflex (LCx), First Obtuse Marginal (OM1), Second Obtuse marginal (OM2), Right CoronaryArtery (RCA), Patent Ductus Arteriosus (PDA), Percutaneous Coronary Intervention (PCI), PCI-LAD, PCI-D1, PCI-D2, PCI-LCx, PCI-OM1, PCI-OM2, PCI-RCA, PCI-PDA, Drug Eluted Stent (DES), Bare Metal Stent (BMS), BMS, Total number of stents, Coronary Artery Bypass Surgery (CABG), Trp post PCI-24, Creatinine-48 post PCI, Stent thrombosis), laboratory findings, history of diabetes (type 1 and 2), Gastroparesis, Erectile dysfunction, Metabolic Syndrome, chronic kidney disease, Chronic Liver Disease, Gestational DM, Diabetic ketoacidosis, hypoglycemia, Hyperosmolar Hyperglycemic Syndrome, Depression, Hypertension, Peripheral Arterial disease, Peripheral Arterial Disease (PAD)- Acute limb ischemia, PAD-Claudication, PAD Critical Limb Ischemia, PAD-Cellulitis, PAD-Lower Limb osteomyelitis, Hemorrhage, Intracranial Hemorrhage, Stroke, Hemorrhagic, Ischemic, Carotid Endarterectomy, carotid Endarterectomy (CEA)-Left, CEA-Right, Carotid stenting, Amputation, Above knee Amputation, Amputation foot, Amputation of Toe, PAD Bypass, PAD intervention, medications.

Study population:

Inclusion criteria: patients with T2DM and established heart disease, such as ischemic heart disease, heart failure, etc. will be included in the study after obtaining the informed consent.

Exclusion criteria: Subjects who do not have T2DM and existing heart disease will be excluded from the registry.

The treating physicians will enter the list of patients attended his clinic to Power Trial. The study investigators will update the list of the patients attended the cardio-metabolic clinic on daily basis and the registry will transfer the information from the Cerner to the registry database. The clinical service has been start from September 15, 2017, and each patient who attended the clinic will be added to the registry.

This registry is prospectively collecting the information from Cerner Clinical Viewer. For future research the investigators who wish to utilize the registry data for their research will have to seek Institutional Review Board (IRB) approval for their research proposal.

Informed Consent Informed consent will be obtained from each patient who will attend the cardiometabolic clinic to allow us to capture his clinical information into the registry database.

Subject Withdrawal/ Withdrawal of Consent If the subjects withdraw his consent, the information about his future follow-up visits in the clinic will not be added to the registry. However, previous data added to the registry will continue to be available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Newly diagnosed heart disease, such as ischemic heart disease, heart failure.

Exclusion Criteria:

* Patients who do not have type 2 diabetes mellitus
* Preexisting heart disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Ten years (15/09/2017 to 31/12/2027)

CONTACTS AND LOCATIONS:
Overall Officials: Jassim Al-Suwaidi, MD, Principal Investigator — Hamad Medical Coorporation
Locations (1):
- Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siscovick DS, Sotoodehnia N, Rea TD, Raghunathan TE, Jouven X, Lemaitre RN. Type 2 diabetes mellitus and the risk of sudden cardiac arrest in the community. Rev Endocr Metab Disord. 2010 Mar;11(1):53-9. doi: 10.1007/s11154-010-9133-5. PMID 20195771
- [Background] Kucharska-Newton AM, Couper DJ, Pankow JS, Prineas RJ, Rea TD, Sotoodehnia N, Chakravarti A, Folsom AR, Siscovick DS, Rosamond WD. Diabetes and the risk of sudden cardiac death, the Atherosclerosis Risk in Communities study. Acta Diabetol. 2010 Dec;47 Suppl 1(Suppl 1):161-8. doi: 10.1007/s00592-009-0157-9. Epub 2009 Oct 24. PMID 19855920
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Shah AD, Langenberg C, Rapsomaniki E, Denaxas S, Pujades-Rodriguez M, Gale CP, Deanfield J, Smeeth L, Timmis A, Hemingway H. Type 2 diabetes and incidence of cardiovascular diseases: a cohort study in 1.9 million people. Lancet Diabetes Endocrinol. 2015 Feb;3(2):105-13. doi: 10.1016/S2213-8587(14)70219-0. Epub 2014 Nov 11. PMID 25466521